CLINICAL TRIAL: NCT06561100
Title: Treatment Optimization of Brain-injured Warfighters: A Prescribed Sub-symptomatic Exercise Treatment
Brief Title: Treatment Optimization of Brain-injured Warfighters
Acronym: (TOBI-SET)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TP210450
Record Dates: First submitted 2024-06-21; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Mild Traumatic Brain Injury
Keywords: Progressive Return to Activity; Warfighter Readiness
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Intervention Model Description: Participants are randomized to one or more study arms and each study arm will be allocated a different intervention.
Who Masked: Outcomes Assessor
Masking Description: Participants will be randomized into either the exercise or stretching condition in a 1:1 fashion. The outcome assessors will be blinded at all times while the intervention specialist (study trainers) will unblind themselves prior to the participants first intervention appointment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sub-symptomatic Adaptable Exercise Treatment (SAET) (Experimental): Participants will attend two in-clinic sessions per week with either a licensed Physical Therapist or Exercise Physiologist and complete three sessions per week independently outside of the clinic. Each session will be 1 hour in duration, 5 days a week for 8 weeks, for a total of 40 hours. Participants will complete a combination of aerobic and resistance training exercises prescribed and adapted to the participant's personal needs based on evaluations by the Physical Therapist and Exercise Physiologist. Exercise will be adjusted to maintain sub-symptomatic levels, meaning that if a participant's neurobehavioral symptoms increase with activity, the intensity and/or exercise will be modified. Furthermore, participants will be asked to fill out an Exercise Habits Questionnaire (EHQ) in order to capture the exercises they are currently doing.
  Interventions: Behavioral: Sub-symptomatic Adaptable Exercise Treatment (SAET)
- Stretching Control Group (SCG) (Active Comparator): Participants will attend two in-clinic sessions per week with either a licensed Physical Therapist or Exercise Physiologist and complete three sessions per week independently outside of the clinic. Each session will be 1 hour in duration, 5 days a week for 8 weeks, for a total of 40 hours. The stretching exercises are designed not to increase heart rate or have excessive head motion consist of static stretching and yoga based movements.
  Interventions: Behavioral: Stretching Control Group (SCG)

INTERVENTIONS:
Behavioral: Sub-symptomatic Adaptable Exercise Treatment (SAET) — Each workout will be structured in a similar format. The first 5 minutes will be devoted to stretching and warm up exercises. Then the next 20 minute segment devoted to light to moderate aerobic exercise. The second 20 minutes of each exercise session will be composed of a series of 5 predetermined exercises that rotate every day. Each workout will have one or two alternatives that the patient can complete either for modification to accommodate a physical limitation or to optimize preference. Resistance training each day will include multi-joint functional movements along with stability work. The last five minutes of the session will include more mobility work, and/or cooling down.
  Arms: Sub-symptomatic Adaptable Exercise Treatment (SAET)
Behavioral: Stretching Control Group (SCG) — Each workout will be 50-60 minutes long and participants are instructed to not do any other type of exercise that may elevate their heart rate. Modifications will be available for stretches that may be too advanced for the individual.
  Arms: Stretching Control Group (SCG)

SUMMARY:
Prescribed sub-symptomatic adaptable exercise treatment (SAET) is a potential solution that promotes recovery needs following a TBI. SAET has been shown to benefit the mind and body in ways that decrease the severity and frequency of mild TBI (mTBI) symptoms. This study aims to validate SAET as an alternative, adaptable treatment or SMs with mTBI that focuses on reducing symptoms, improving mental health, increasing physiological functioning, and ultimately returning to duty.

The objective of this study is to develop a prescribed exercise treatment program for warfighters with mTBI that can be personalized for SM's needs (i.e., medical and occupational) and is adaptable to various clinical resources (e.g., forward operating bases, rural clinics, and mTBI specialty programs). The key question raised by this study is whether SAET is more effective than a stretching control group (SCG) in reducing neurobehavioral symptoms among SMs with persistent complaints following a mTBI.

DETAILED DESCRIPTION:
The study will be a randomized clinical trial among active duty service members (SMs) with persistent cognitive complaints following mTBI, comparing a prescribed sub-symptomatic adaptable exercise treatment (SAET) to an active stretching control group (SCG). SAET's overall effectiveness will be assessed by neurobehavioral symptom resolution. Additional exploratory aims will include cognitive performance, physiological adaptation and locomotion as well as functional changes in military performance. These items will be addressed in the following aims.

Primary Aim:

To determine whether SAET is more effective than the control condition in reducing neurobehavioral symptoms among SMs with persistent complaints following mTBI. Hypothesis 1: There will be a greater reduction in the Neurobehavioral Symptoms Inventory (NSI) from pre- to post-SAET compared to the control condition. A similar finding will continue from immediate to 3 month post-SAET.

Secondary Aims:

Sub-aim 1 Cognitive Status: To determine if SAET is effective at improving cognitive impairment among SMs with persistent complaints from mTBI. Sub-hypothesis 1: There will be a greater decrease in the Global Deficit Scores (GDS; an overall measure of cognitive impairment) post SAET in comparison to the control condition.

Sub-aim 2 Physiological Adaptation: To measure physiological adaptation associated with SAET compared to the control condition. Sub-hypothesis 2: SAET will be associated with improved cerebrovascular blood flow regulation, as measured by Transcranial Doppler and improved cardiovascular function, as measured by changes in heart rate variability (HRV) and estimated maximal oxygen consumption (est. VO2 max) compared to the control condition.

Sub-aim 3 Warfighter Performance: To determine if SAET participants will have improved locomotion and a higher level of occupational performance compared to the control condition. Sub-hypothesis 3: SAET participants will have improved locomotion and physical performance (based on the Marine Corps Combat Fitness Test(CFT)) and higher ratings of occupational performance (based on supervisor ratings on the Checklist of Military Activities of Daily Living [M-ADL]) after completion of treatment and 3 months post-treatment compared to the control condition.

ELIGIBILITY:
Inclusion Criteria:

* Active duty, male or female, ages 18 to 55
* History of at least one mTBI sustained more than 1 month ago
* Service members (SMs) with ongoing symptoms

Exclusion Criteria:

* SMs who sustained a TBI of any severity within 1 month of enrollment
* History of moderate, severe, or penetrating TBI
* Current substance use disorder
* History of a neurological disease (e.g., multiple sclerosis, cerebral vascular accident, brain tumor, neurodegenerative disease, or neuro-motor disorder)
* An acute orthopedic injury that limits the capacity to complete study procedures

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Neurobehavioral Symptom Change | 6 Months
  Change in the Neurobehavioral Symptoms Inventory (NSI) from pre- to post-SAET.
  Neurobehavioral symptoms will be assessed using the Neurobehavioral Symptom Inventory (NSI) which captures multiple neurobehavioral symptoms including cognitive, somatosensory, vestibular, and affective. Furthermore, this 22 item self-report questionnaire is well validated in research studies on TBI in military populations, it has known reliability and validity, as well as guidelines for assessment of change.

SECONDARY OUTCOMES:
Cognitive Impairment Change | 6 Months
  There will be a change in the Global Deficit Scores (GDS; an overall measure of cognitive impairment) post intervention.
Maximal oxygen consumption | 6 Months
  We will measure cardiovascular fitness levels by administering an estimated maximal Oxygen consumption (est. VO2 max) test. Fitness levels will be determined based on VO2 percentage and categorized by very low, low, fair, good, excellent, or superior fitness level.
Warfighter readiness based on Combat Fitness Test | 6 Months
  We will measure changes in locomotion, physical performance (based on the Marine Corps Combat Fitness Test (CFT)), after completion of treatment and 3 months post-treatment. A CFT classification score ranging from 1st class through 3rd class or failed, will be given based on their performance.
Change in level of occupational performance | 6 months
  Ratings of occupational performance by a direct supervisor using a modified Checklist of Military Activities of Daily Living (M-ADL).

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Bailie, Phd, Principal Investigator — Traumatic Brain Injury Center of Excellence (TBICoE)
Locations (1):
- Intrepid Spirit Center, Camp Pendleton, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All surveys, questionnaires, and other instruments will be aligned with Federal Interagency Traumatic Brain Injury Research Informatics System (FITBIR) when possible. FITBIR is a central repository for data from TBI studies built by the National Institute of Health and the Department of Defense.
Supporting Information: Study Protocol
Time Frame: The data will be uploaded and available after study completion. IT is unsure for how long the data is available but FITBIR's confidentiality certificate is approved till 16 July 2032.
Access Criteria: In order to access FITBIR's data repository, an account has to be created in which access is then granted to the user.
URL: https://fitbir.nih.gov/

DOCUMENTS (2):
  • Study Protocol (2024-01-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT06561100/Prot_000.pdf
  • Informed Consent Form (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT06561100/ICF_001.pdf